CLINICAL TRIAL: NCT05779098
Title: A Machine Learning Architecture to Predict Post-Hepatectomy Liver Failure Using Liver Regeneration Biomarkers and Time-Phased Data
Acronym: PHLF predictio
Status: Completed | Type: Observational
Sponsor: Shen Feng (Other)
Collaborators: Shanghai 10th People's Hospital (Other); Jinling Hospital, China (Other)
Responsible Party: Sponsor-Investigator, Shen Feng, Dean of Clinical Research Institute of Eastern Hepatobiliary Surgery Hospital, Eastern Hepatobiliary Surgery Hospital
Organization: Eastern Hepatobiliary Surgery Hospital (Other)
Other Study IDs: 1312871874
Record Dates: First submitted 2023-03-09; First posted 2023-03-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Liver Failure After Operative Procedure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Extensive hepatectomy

SUMMARY:
Post-hepatectomy liver failure (PHLF) is the leading cause of morbidity and mortality following major hepatectomy. Existing prediction models fail to capture the dynamic liver regeneration and perioperative changes, limiting their predictive accuracy. We aimed to develop a machine learning (ML) modelling system (PILOT architecture) integrating liver regeneration biomarkers with time-phased perioperative clinical data to accurately predict PHLF risk.

ELIGIBILITY:
Inclusion Criteria:

Extensive hepatectomy in our hospital（≥ three Hepatic segment）

Exclusion Criteria:

Serious basic diseases Intolerable surgery Refuse to perform ICG test before operation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Extensive Hepatology in our hospital
Sampling Method: Non-Probability Sample
Enrollment: 1071 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Postoperative liver failure | 1-5 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Hepatobiliary and Pancreatic Surgery, Tenth People's Hospital of Tongji University, School of Medicine, Tongji University, Shanghai, China, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shen H, Yuan T, Si A, Shen Y, Liu J, Jin L, Xie Z, Zhang H, Wei W, Dai Y, Jiang T, He C, Zhang S, Hu Y, Huang S, Yang Z, Chen Y, Zhang X, Shen F, Qi X, Li J. Liver regeneration-associated machine learning architecture integrating time-phased predictions for post-hepatectomy liver failure. EClinicalMedicine. 2025 Nov 28;90:103661. doi: 10.1016/j.eclinm.2025.103661. eCollection 2025 Dec. PMID 41399475